CLINICAL TRIAL: NCT03222557
Title: Electroacupuncture for Postoperative Ileus After Laparoscopic Surgery for Mid and Low Rectal Cancer: A Prospective, Randomized, Sham-controlled Trial
Brief Title: Electroacupuncture for Postoperative Ileus After Laparoscopic Surgery for Mid and Low Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor of Surgery, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CREC Ref. No.: 2017.010-T
Record Dates: First submitted 2017-07-14; First posted 2017-07-19 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Postoperative Ileus; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The acupuncturist is the only individual who is aware of the treatment allocation; the patients randomized to the EA/SA groups and the outcome assessor are blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (EA) (Experimental): Bilateral acupoints relevant to the treatment of abdominal pain, abdominal distension, and constipation, including Zusanli (stomach meridian ST-36), Sanyinjiao (spleen meridian SP-6), Hegu (large intestine meridian LI-4), and Zhigou (triple energizer meridian TE-6), will be used. Electric stimulation at a frequency of 50 Hz will be employed to the needles
  Interventions: Procedure: Electroacupuncture; Device: Electroacupuncture
- Sham Acupuncture (SA) (Sham Comparator): Sterile blunt-tip needles will be placed (without skin penetration) 20 mm away from the acupoints. The needle will be first inserted through a sterile plastic tube mounted on a foam block, and then pressed on the skin. The foam block compresses to give the impression that the needle is penetrating the skin, thus providing a SA effect. 'Pseudostimulation' will be given by deliberately connecting the needle to the incorrect output socket of the electroacupuncture device, thus there will be no flow of electric current.
  Interventions: Procedure: Sham Acupuncture; Device: Sham Acupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Refer to arm description
  Other Names: EA
  Arms: Electroacupuncture (EA)
Procedure: Sham Acupuncture — Refer to arm description
  Other Names: SA
  Arms: Sham Acupuncture (SA)
Device: Electroacupuncture — Refer to arm description
  Other Names: EA
  Arms: Electroacupuncture (EA)
Device: Sham Acupuncture — Refer to arm description
  Other Names: SA
  Arms: Sham Acupuncture (SA)

SUMMARY:
This is a prospective, randomized, sham-controlled, superiority trial that aimed to investigate the efficacy of electroacupuncture (EA) in reducing the duration of postoperative ileus and hospital stay after laparoscopic total mesorectal excision or abdominoperineal resection for rectal cancer.

DETAILED DESCRIPTION:
Background: Postoperative ileus (POI) remains a significant problem after colorectal surgery that adversely influences patients' recovery and prolongs hospital stay. The investigators' previous study demonstrated that electroacupuncture (EA) at Zusanli, Sanyinjiao, Hegu, and Zhigou reduces the duration of POI and hospital stay after laparoscopic resection of colonic and upper rectal cancer (Ng et al. Gastroenterology 2013; 144: 307-313). However, patients with mid/low rectal cancer undergoing laparoscopic sphincter-preserving total mesorectal excision (TME) or abdominoperineal resection (APR) were excluded. These complicated cases are apparently more likely to develop prolonged ileus and morbidity after surgery.

Objectives: To investigate the efficacy of EA in reducing the duration of POI and hospital stay after laparoscopic TME or APR for rectal cancer.

Hypothesis: Rectal cancer patients undergoing laparoscopic TME or APR within a fast-track perioperative program who receive EA will have shorter duration of POI and hospital stay when compared with those who receive sham acupuncture (SA).

Design: Prospective, randomized, sham-controlled, superiority trial.

Subjects: One hundred and sixty four consecutive patients with mid/low rectal cancer undergoing laparoscopic surgery without the need of conversion will be recruited. All patients will follow a standard perioperative fast-track program.

Interventions: Patients will be randomly allocated to receive either EA or SA. Bilateral acupoints including Zusanli, Sanyinjiao, Hegu, and Zhigou will be used. The acupuncturist is the only individual who is aware of the treatment allocation; the patients randomized to the EA/SA groups and the outcome assessor are blinded to the treatment allocation. The patients will undergo one session of EA daily from day 1 till day 4, or until the time when the primary outcome has occurred, whichever is earlier.

Outcome measures: Primary outcome: a composite endpoint of time to recovery of upper and lower gastrointestinal function (GI-2). Secondary outcomes: time to discharge order written, length of hospital stay, postoperative pain scores and analgesic requirement, and postoperative 30-day morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients (aged between 18 and 80) with mid/low rectal cancer (adenocarcinoma in the rectum of which the lowest margin of the tumor is located within 12 cm of the anal verge as measured by rigid sigmoidoscopy) undergoing laparoscopic sphincter-preserving TME or APR without the need of conversion
* American Society of Anesthesiologists grading I-III
* Informed consent available

Exclusion Criteria:

* Patients with previous experience of acupuncture
* Those undergoing simultaneous laparoscopic resection of rectal cancer and other coexisting intraabdominal diseases
* Those undergoing laparoscopic resection of rectal cancer with en bloc resection of surrounding organs
* Those who developed intraoperative problems or complications (e.g. bleeding, tumor perforation) that required conversion
* Those undergoing emergency surgery
* Those with previous history of midline laparotomy
* Those with evidence of peritoneal carcinomatosis
* Those who are expected to receive epidural anesthesia or analgesia
* Those with cardiac pacemaker
* Those who are pregnant
* Those who are allergic to the acupuncture needles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
GI-2 recovery | Up to 10 days
  A composite assessment that measured upper (first tolerance of solid food) and lower (first bowel movement) GI tract recovery, with time to achieve GI-2 recovery based on the last event to occur

SECONDARY OUTCOMES:
Time of first passing flatus | Up to 10 days
Length of hospital stay | Up to 1 month
Pain scores on the first 3 postoperative days | Up to postoperative day 3
  On visual analog scale (from 0 which implies no pain at all, to 10 which implies the worst pain imaginable)
Postoperative analgesic requirement | Up to 1 month
Short-term morbidity | Up to 1 month
  Defined by the Clavien-Dindo classification of surgical complications
Adverse events related to EA/SA | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No